CLINICAL TRIAL: NCT02957968
Title: T-Cell Immune Checkpoint Inhibition Plus Hypomethylation for Locally Advanced HER2-Negative Breast Cancer - A Phase 2 Neoadjuvant Window Trial of Pembrolizumab and Decitabine Followed by Standard Neoadjuvant Chemotherapy
Brief Title: Neoadjuvant Pembrolizumab + Decitabine Followed by Std Neoadj Chemo for Locally Advanced HER2- Breast Ca
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15-11083; NCI-2016-01980 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA016059 (NIH)
Record Dates: First submitted 2016-11-03; First posted 2016-11-08 (Estimated); Results first posted 2023-11-09 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Breast Adenocarcinoma; Estrogen Receptor- Negative Breast Cancer; Estrogen Receptor-positive Breast Cancer; HER2/Neu Negative; Invasive Breast Carcinoma; Progesterone Receptor Negative; Progesterone Receptor Positive Tumor; Stage II Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Triple-negative Breast Carcinoma
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Paclitaxel; Albumin-Bound Paclitaxel; Carboplatin; Decitabine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Triple Negative Breast Cancer (TNBC) (Experimental): Triple Negative Breast Cancer (Cohort A): Decitabine IV over 60 minutes on 4 days and pembrolizumab IV over 30 minutes on days 8 and 22. Four cycles of dose-dense doxorubicin and cyclophosphamide (AC), followed by 12 doses of weekly paclitaxel and carboplatin.
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Carboplatin; Drug: Decitabine; Drug: Pembrolizumab
- Cohort B: HER2-negative hormone receptor-positive tumors (Experimental): HER2-negative hormone receptor-positive tumors (Cohort B): Decitabine IV over 60 minutes on 4 days and pembrolizumab IV over 30 minutes on days 8 and 22. Four cycles of dose-dense doxorubicin and cyclophosphamide (AC), followed by 12 doses of weekly paclitaxel.
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Decitabine; Drug: Pembrolizumab
- Cohort A2: Triple Negative Breast Cancer (TNBC) with Extended Pembrolizumab (Experimental): Triple Negative Breast Cancer (Cohort A2). Decitabine IV over 60 minutes on 4 days and pembrolizumab IV over 30 minutes on days 8 and 22. Four cycles of dose-dense doxorubicin and cyclophosphamide (AC), followed by 12 doses of weekly paclitaxel and carboplatin, and pembrolizumab every 3 weeks.
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Carboplatin; Drug: Decitabine; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Doxorubicin — 60 mg/m2 once every 2 weeks for 4 cycles.
  Other Names: Adriamycin; Rubex
Drug: Cyclophosphamide — cyclophosphamide 600 mg/m2 (AC) once every 2 weeks for 4 cycles.
  Other Names: Cytoxan; Neosar
Drug: Paclitaxel — Paclitaxel 80 mg/m2 IV once weekly for 12 weeks.
  Other Names: Taxol; Onxol; Abraxane
Drug: Carboplatin — carboplatin IV 1.5 area under curve (AUC) once weekly for 12 weeks.
  Other Names: Paraplatin
  Arms: Cohort A2: Triple Negative Breast Cancer (TNBC) with Extended Pembrolizumab; Cohort A: Triple Negative Breast Cancer (TNBC)
Drug: Decitabine — Given IV
  Other Names: Dacogen; Deoxyazacytidine; Dezocitidine
Drug: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab

SUMMARY:
This study is a 2-cohort, open-label, multicenter, phase 2 study of a short course of immunotherapy consisting of sequential decitabine followed by pembrolizumab administered prior to a standard neoadjuvant chemotherapy regimen for patients with locally advanced HER2-negative breast cancer. The primary efficacy objective is to determine if the immunotherapy increases the presence and percentage of tumor and/or stromal area of infiltrating lymphocytes prior to initiation of standard neoadjuvant chemotherapy. At enrollment, patients will be assigned to one of 2 cohorts based on hormone receptor status.

* Cohort A - patients with HER2-negative, hormone receptor-negative breast cancer (defined as both ER and PgR with < 10% positive staining on IHC) Note: before beginning standard neoadjuvant chemotherapy, patients in Cohort A may be reassigned to Cohort A2 to receive extended pembrolizumab as part of new standard neoadjuvant and postoperative adjuvant therapy.
* Cohort B - patients with HER2-negative, hormone receptor-positive breast cancer (defined as either ER or PgR with ≥ 10% positive staining on IHC)

DETAILED DESCRIPTION:
Both cohorts will receive the identical doses and treatment schedules of decitabine and pembrolizumab followed by a standard neoadjuvant chemotherapy regimen. Both cohorts will receive 4 cycles of AC and 12 doses of weekly paclitaxel or Nab-paclitaxel. Paclitaxel or Nab-paclitaxel will be combined with carboplatin for Cohorts A and A2 (TNBC). The sequence of the 2 regimens will be at the discretion of the treating medical oncologist following the safety lead-in phase. For the primary endpoint, Cohorts A and A2 will be evaluated together, separate from Cohort B.

ELIGIBILITY:
Inclusion Criteria:

* Invasive adenocarcinoma of the breast diagnosed by core needle biopsy
* Breast cancer determined to be HER2-negative per current American Society of Clinical Oncologists/College of American Pathologists (ASCO/CAP) human epidermal growth factor receptor 2 (HER2) Guidelines (If IHC was performed, IHC 0 or 1+; if fluorescence in situ hybridization (FISH) or other in situ hybridization test, dual probe HER2/Chromosome 17 Centromere (CEP17) ratio < 2.0 with an average HER2 copy number < 4.0 signals/cell)
* Breast cancer determined to be hormone receptor-positive or hormone receptor-negative defined as follows:

  * Hormone receptor-positive: ≥ 10% staining by IHC for either estrogen receptor (ER) or progesterone receptor (PgR)
  * Hormone receptor-negative: < 10% staining by IHC for both ER and PgR
* Locally advanced breast cancer defined as any of the following per American Joint Committee on Cancer (AJCC) Staging Criteria:

  * T2 based on tumor measurements by physical examination or imaging and with clinically positive regional lymph nodes (cN1 or cN2), irrespective of hormone receptor status
  * Hormone receptor-negative breast cancer patients with tumor size of 3-5 cm measured by physical examination or imaging with clinically negative regional lymph nodes (cN0)
  * Any T3 based on tumor measurements by physical examination or imaging
  * Any T4 (including inflammatory breast cancer), irrespective of hormone receptor status
* Ipsilateral axillary lymph nodes must be evaluated by MRI or ultrasound within 12 weeks prior to study registration to determine clinical nodal status. If imaging is suspicious or abnormal, a fine needle aspiration (FNA) or core biopsy of the questionable node(s) on imaging is required. Nodal status should be classified according to the following criteria:

  * Nodal status - negative

    * Imaging of the axilla is negative; OR
    * Imaging of the axilla is suspicious or abnormal AND FNA or core biopsy is negative.
  * Nodal status - positive

    * FNA or core biopsy of node(s) is cytologically or histologically suspicious or positive
* Breast imaging performed prior to study registration as follows:
* Ipsilateral breast - within 12 weeks
* Contralateral breast - within 24 weeks
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate bone marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1,500/mm3
  * Platelet count ≥ 100,000/mm3
  * Hemoglobin ≥ 10.0 g/dL
* Adequate renal function as defined below:
* Serum creatinine ≤ upper limit of normal (ULN) for the lab or a calculated creatinine clearance ≥ 60 mL/min
* Adequate hepatic function as defined below:

  * Total bilirubin ≤ ULN for the laboratory
  * Aspartate aminotransferase (AST) ≤ 1.5 x ULN for the laboratory
  * Alanine aminotransferase (ALT) ≤ 1.5 x ULN for the laboratory
  * Alkaline phosphatase (ALP) ≤ 2.5 x ULN for the laboratory Note: If ALP is > 1.5 x ULN, imaging to rule out bone and liver metastasis is required.
* Left ventricular ejection fraction (LVEF) assessment (ie, 2-D echocardiogram or multigated acquisition (MUGA) scan) performed within 12 weeks prior to study registration indicates an LVEF ≥ 50% regardless of the cardiac imaging facility's lower limit of normal
* Women who are not postmenopausal or have not undergone hysterectomy must have a documented negative serum pregnancy test within 72 hours prior to initiating study treatment.

Note: Postmenopausal is defined as any of the following:

* Age ≥ 60 years
* Age < 60 years and amenorrheic for at least 1 year with follicle-stimulating hormone (FSH) and plasma estradiol levels in the postmenopausal range
* Bilateral oophorectomy

  * A female patient who is a woman of child-bearing potential (WCBP) and a male patient with a partner who is a WCBP must agree to use a medically accepted method for preventing pregnancy for the duration of immunotherapy and neoadjuvant chemotherapy and until after completion of breast surgery or, for patients who do not receive neoadjuvant chemotherapy, for a minimum of 6 months following the last dose of pembrolizumab or decitabine
  * Ability to understand and willingness to sign the consent form

Exclusion Criteria:

* Breast cancer treatment for the currently diagnosed breast cancer including radiation therapy, chemotherapy, targeted therapy, or endocrine therapy prior to study registration
* Administration of a live vaccine within 30 days prior to initiating study treatment Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are permitted; however, intranasal influenza vaccines (eg, Flu-Mist) are live attenuated vaccines, and are not allowed.
* Administration of a monoclonal antibody within 4 weeks prior to initiating study treatment or has not recovered (ie, ≤ grade 1 or at baseline) from adverse events (AEs) due to a monoclonal antibody administered more than 4 weeks earlier
* Administration of any investigational agent within 4 weeks prior to initiating study treatment
* Evidence of metastatic disease that is extensive enough to preclude consideration of subsequent definitive surgery for the primary tumor
* History of ipsilateral invasive breast cancer or ipsilateral ductal carcinoma in situ (DCIS) Note: Patients with history of ipsilateral lobular carcinoma in situ (LCIS) are eligible.
* History of solid organ or allogeneic stem cell transplant
* Previous therapy for any malignancy with an anthracycline or taxane for Cohorts A and B and carboplatin for Cohort A
* Cardiac disease that would preclude administration of the drugs included in the study treatment regimen including, but not limited to:

  * Angina pectoris that requires the current use of anti-anginal medication
  * Ventricular arrhythmias except for benign premature ventricular contractions
  * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
  * Conduction abnormality requiring a pacemaker
  * Valvular disease with documented compromise in cardiac function; and symptomatic pericarditis
* Nervous system disorder (ie, paresthesia, peripheral motor neuropathy, or peripheral sensory neuropathy) ≥ grade 2, per CTCAE v5.0
* Administration of or condition requiring administration of systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to initiating study treatment Exception: Patients with conditions that can be managed with steroids equivalent to or less than an oral prednisone dose of 10 mg daily would not be excluded from the study.
* Previous therapy for this cancer with an anti-anti-programmed death-1 (PD-1), anti-PD-L1, anti-PD-L2 agent, or any other immunomodulatory agent
* Known or presumed hypersensitivity to decitabine or pembrolizumab (or any of their excipients)
* Diagnosed immunodeficiency, eg, human immunodeficiency virus (HIV)
* Active autoimmune disease requiring systemic treatment within the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs) or a documented history of clinically severe autoimmune disease or a syndrome that requires systemic steroids or immunosuppressive agents Note: Patients with the conditions or medical history listed below are NOT excluded from this study.

  * Vitiligo
  * Resolved childhood asthma/atopy
  * Requirement for intermittent use of bronchodilators or local steroid injections or topical steroids
  * Hypothyroidism stable on hormone replacement
  * Sjogren's Syndrome
* Known history or evidence of interstitial lung disease or active, non-infectious pneumonitis
* Known history of active bacillus tuberculosis (TB)
* Active infection requiring systemic therapy
* Known active Hepatitis B or C
* Pregnancy or breastfeeding
* Diagnosis or treatment for another malignancy within 5 years prior to study registration, with the following exceptions: complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, any in situ malignancy, and low-risk prostate cancer after curative therapy
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Harry D. Bear, M.D., Ph.D., Principal Investigator — Massey Cancer Center
Locations (4):
- United States (4):
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Background] Bear HD, Deng X, Bandyopadhyay D, Idowu M, Jenkins TM, Kmieciak M, Williams M, Archer G, Gwaltney L, Dillon P, Flora D, Stover D, Poklepovic AS, Hackney M, Ross M, Vachhani H, Louie R, McGuire KP, Grover A, Rahman T, Hendrix A. T-cell immune checkpoint inhibition plus hypomethylation for locally advanced HER2-negative breast cancer: a phase 2 neoadjuvant window trial of decitabine and pembrolizumab followed by standard neoadjuvant chemotherapy. J Immunother Cancer. 2025 Feb 27;13(2):e010294. doi: 10.1136/jitc-2024-010294. PMID 40021215

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Triple Negative Breast Cancer (TNBC): Triple Negative Breast Cancer (Cohort A): Decitabine IV over 60 minutes on 4 days and pembrolizumab IV over 30 minutes on days 8 and 22. Four cycles of dose-dense doxorubicin and cyclophosphamide (AC), followed by 12 doses of weekly paclitaxel and carboplatin.
  Doxorubicin: 60 mg/m2 once every 2 weeks for 4 cycles.
  Cyclophosphamide: cyclophosphamide 600 mg/m2 (AC) once every 2 weeks for 4 cycles.
  Paclitaxel: Paclitaxel 80 mg/m2 IV once weekly for 12 weeks.
  Carboplatin: carboplatin IV area under curve ( AUC) 1.5 once weekly for 12 weeks.
  Decitabine: Given IV
  Pembrolizumab: Given IV
- Cohort B: HER2-negative Hormone Receptor-positive Tumors: Human epidermal growth factor receptor 2 (HER2)-negative hormone receptor-positive tumors (Cohort B): Decitabine IV over 60 minutes on 4 days and pembrolizumab IV over 30 minutes on days 8 and 22. Four cycles of dose-dense doxorubicin and cyclophosphamide (AC), followed by 12 doses of weekly paclitaxel.
  Doxorubicin: 60 mg/m2 once every 2 weeks for 4 cycles.
  Cyclophosphamide: cyclophosphamide 600 mg/m2 (AC) once every 2 weeks for 4 cycles.
  Paclitaxel: Paclitaxel 80 mg/m2 IV once weekly for 12 weeks.
  Decitabine: Given IV
  Pembrolizumab: Given IV
- Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab: Triple Negative Breast Cancer (Cohort A2). Decitabine IV over 60 minutes on 4 days and pembrolizumab IV over 30 minutes on days 8 and 22. Four cycles of dose-dense doxorubicin and cyclophosphamide (AC), followed by 12 doses of weekly paclitaxel and carboplatin, and pembrolizumab every 3 weeks.
  Doxorubicin: 60 mg/m2 once every 2 weeks for 4 cycles.
  Cyclophosphamide: cyclophosphamide 600 mg/m2 (AC) once every 2 weeks for 4 cycles.
  Paclitaxel: Paclitaxel 80 mg/m2 IV once weekly for 12 weeks.
  Carboplatin: carboplatin AUC 1.5 once weekly for 12 weeks.
  Decitabine: Given IV
  Pembrolizumab: Given IV
Period: Overall Study
Arm/Group | Cohort A: Triple Negative Breast Cancer (TNBC) | Cohort B: HER2-negative Hormone Receptor-positive Tumors | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab
Started | 21 | 18 | 7
Completed | 17 | 14 | 6
Not Completed | 4 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort A: Triple Negative Breast Cancer (TNBC): Triple Negative Breast Cancer (Cohort A): Decitabine IV over 60 minutes on 4 days and pembrolizumab IV over 30 minutes on days 8 and 22. Four cycles of dose-dense doxorubicin and cyclophosphamide (AC), followed by 12 doses of weekly paclitaxel and carboplatin.
  Doxorubicin: 60 mg/m2 once every 2 weeks for 4 cycles.
  Cyclophosphamide: cyclophosphamide 600 mg/m2 (AC) once every 2 weeks for 4 cycles.
  Paclitaxel: Paclitaxel 80 mg/m2 IV once weekly for 12 weeks.
  Carboplatin: carboplatin AUC 1.5 once weekly for 12 weeks.
  Decitabine: Given IV
  Pembrolizumab: Given IV
- Total: Total of all reporting groups
Arm/Group | Cohort A: Triple Negative Breast Cancer (TNBC) | Cohort B: HER2-negative Hormone Receptor-positive Tumors | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab | Total
Number analyzed (Participants) | 21 | 18 | 7 | 46
Age, Continuous [Median (Full Range); unit: Years] | 56 [35 to 72] | 54 [28 to 70] | 55 [28 to 65] | 54.5 [28 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 7 | 46
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 21 | 17 | 7 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 1 | 13
  White | 15 | 12 | 6 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 18 | 7 | 46

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Increase in Tumor and Stroma With Infiltrating Lymphocytes (TIL) From Baseline Pre-treatment Biopsy to Post-immunotherapy Biopsy Following Administration of Decitabine Followed by Pembrolizumab.
Description: To determine and quantify if treatment with neoadjuvant decitabine followed by pembrolizumab increases lymphocyte infiltration into tumor and/or stroma in patients with locally advanced, HER2-negative breast cancer.
Time Frame: Baseline pre-treatment biopsy to post-immunotherapy biopsy following administration of decitabine followed by pembrolizumab, 3-7 day window after Day 22 medication administration, about one month
Measure: Mean (Standard Deviation); unit: % of stromal area occupied by TIL
Arm/Group | Cohort A: Triple Negative Breast Cancer (TNBC) | Cohort B: HER2-negative Hormone Receptor-positive Tumors | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab
Number analyzed (Participants) | 17 | 14 | 6
% of stromal area occupied by TIL
  Baseline | 27.35 (17.69) | 17.50 (9.95) | 25.83 (12.01)
  Post Treatment | 35.00 (21.43) | 23.57 (12.00) | 32.50 (11.73)
  Absolute Change Value | 7.65 (15.12) | 6.07 (8.13) | 6.67 (12.11)

2. Secondary Outcome: Number of Adverse Events (AEs) Reported During and After Immune Treatment (ie, Decitabine and Pembrolizumab)
Description: Using criteria in the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0), all adverse events (AEs) regardless of grade or attribution, will be captured from the beginning of study treatment (initiation of decitabine) until initiation of standard neoadjuvant chemotherapy.
  For patients who do not initiate pembrolizumab, all AEs will be captured until 30 days following the last dose of decitabine or until another cancer treatment is initiated, whichever occurs first.For patients who initiate pembrolizumab, immune related adverse events (irAEs) (clinically significant and non-clinically significant) will be captured from the initiation of pembrolizumab through the end of the 30- day post-surgery (or post-treatment, for those who don't have surgery) follow-up period and at a 12-month follow-up time point.
Time Frame: Time of study registration until 30 days following the end of administration of decitabine and pembrolizumab, or until another cancer treatment was initiated, or 30 days following surgery, 12- months.
Measure: Number; unit: Adverse Events Reported
Arm/Group | Cohort A: Triple Negative Breast Cancer (TNBC) | Cohort B: HER2-negative Hormone Receptor-positive Tumors | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab
Number analyzed (Participants) | 21 | 18 | 7
Adverse Events Reported | 215 | 151 | 98

3. Secondary Outcome: Number of Patients Meeting Criteria for Lymphocyte-predominant Breast Cancer (LPBC) Following Treatment With Decitabine and Pembrolizumab
Description: To determine if the study treatment increases the proportion of tumors with ≥ 60% tumor or stromal area infiltrated with lymphocytes (ie, LPBC). The percentage of patients meeting criteria for LPBC following treatment with decitabine and pembrolizumab compared to the percentage before treatment (LPBC is defined as breast cancer with ≥ 60% intratumoral or stromal area with infiltrating lymphocytes.)
Time Frame: Assessed at end of administration of decitabine and pembrolizumab Day- Window of time Days 25-29
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Triple Negative Breast Cancer (TNBC) | Cohort B: HER2-negative Hormone Receptor-positive Tumors | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab
Number analyzed (Participants) | 17 | 14 | 6
Participants | 3 | 0 | 0

4. Secondary Outcome: Number of Patients With Pathologic Complete Response (pCR) in the Breast and Post-therapy Lymph Nodes.
Description: To determine the rate of pCR in the breast and lymph nodes (pCR breast and nodes). The number of patients with pCR in the breast and post-therapy lymph nodes defined as the absence of any invasive cancer in the resected breast specimen and absence of cancer on H&E evaluation of all resected lymph nodes following completion of neoadjuvant therapy (ypT0/is; ypN0).
Time Frame: End of administration of decitabine and pembrolizumab Day- Window of time Days 25-29, or 30 days following surgery
Population: All participants in trial either did not have surgery performed, or did not have a suitable biopsy, therefore pathological response could not be assessed for all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Triple Negative Breast Cancer (TNBC) | Cohort B: HER2-negative Hormone Receptor-positive Tumors | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab
Number analyzed (Participants) | 20 | 16 | 7
Participants | 10 | 3 | 1

5. Secondary Outcome: Number of Patients With no or Minimal Residual Disease in the Resected Breast and Axillary Specimen.
Description: To determine the rate of Residual Cancer Burden (RCB) Index value of 0-1 following all neoadjuvant therapy. The number of patients with no (0) or (i) minimal residual disease in the resected breast and axillary specimen defined as RCB Index value 0 or i (Arabic numeral).
Time Frame: End of therapy surgery
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Triple Negative Breast Cancer (TNBC) | Cohort B: HER2-negative Hormone Receptor-positive Tumors | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab
Number analyzed (Participants) | 13 | 5 | 2
Participants
  0 (no MRD) | 10 | 3 | 1
  i (MRD present) | 3 | 2 | 1

6. Secondary Outcome: The Number of Patients With Clinical Complete Response (cCR)
Description: To determine the rate of clinical complete response in the breast and lymph nodes (cCR breast and nodes) following all neoadjuvant therapy. The proportion of patients with cCR defined as the absence of tumor based on physical examination of the breast and nodes following completion of all neoadjuvant therapy.
Time Frame: End of therapy surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Triple Negative Breast Cancer (TNBC) | Cohort B: HER2-negative Hormone Receptor-positive Tumors | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab
Number analyzed (Participants) | 20 | 16 | 7
Participants
  cCR=No | 6 | 8 | 5
  cCR=Yes | 14 | 8 | 2

7. Secondary Outcome: Enumeration of T Cells and Immune Cell Subsets
Description: To characterize the alteration of T lymphocyte and other host cell infiltration and immune response gene signatures in breast cancers resulting from treatment with decitabine and pembrolizumab. Enumeration of T cells and immune cell subsets, including cluster of differentiation 8 (CD8)+ cytotoxic T cells, cluster of differentiation 4 (CD4)+ helper T cells, FOXP3+ regulatory T Cells, cluster of differentiation 20 (CD20)+ B cells, and MDSC in the tumor sample procured by core needle biopsy following completion of sequential decitabine followed by pembrolizumab compared to the number of these cells in tumor samples procured at baseline.
Time Frame: Assessed at end of administration of decitabine and pembrolizumab Day- Window of time Days 25-29
Reporting Status: Not Posted, anticipated posting 2026-03

8. Secondary Outcome: Evaluation of Expression of Protein Programmed Death-Ligand 1 (PD-L1) Within Tumor, Stroma, and Infiltrating Immune Cells Combined, at Baseline and Following Immunotherapy.
Description: To evaluate the correlation of pre-existing and post-immunotherapy immune response signatures with response to neoadjuvant chemotherapy. The number of PD-L1 positive cells (including tumor cells, lymphocytes, and macrophages) divided by the total number of tumor cells (PD-L1 positive or negative) in an area.
Time Frame: Assessed at end of administration of decitabine and pembrolizumab Day- Window of time Days 25-29
Population: Not all participants had surgery performed, therefore response could not be assessed for all patients (3/36). Specimen issues limited number who could have PD-L1 assessments to 37/46
Measure: Mean (Standard Deviation); unit: Number of PD-L1 positive cells
Arm/Group | Cohort A: Triple Negative Breast Cancer (TNBC) | Cohort B: HER2-negative Hormone Receptor-positive Tumors | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab
Number analyzed (Participants) | 17 | 14 | 6
Number of PD-L1 positive cells
  Baseline (Bx 1) | 31.00 (29.63) | 13.07 (17.22) | 22.50 (23.36)
  Post Immunotherapy | 50.00 (34.73) | 29.07 (28.15) | 35.50 (26.04)
  Change (Bx2-Bx1) | 19.00 (24.27) | 16.00 (28.15) | 13.00 (17.12)

9. Secondary Outcome: Change of Intensity of Programmed Death-Ligand 1 (PD-L1) Expression by Assay as it Relates to Pathologic Complete Response (pCR) Rates From Chemotherapy
Description: Combined positive score (CPS) is calculated by the number of PD-L1 positive cells, including tumor cells, lymphocytes, and macrophages divided by the total number of viable tumor cells multiplied by 100 (n>100 is possible). The point biserial correlation coefficient (RPB) was calculated to quantify the association between the binary factor (BFA) pCR,and continuous factor PD-L1-CPS. The two PD-L1-cps variables (BX2_PD-L1_cps, Change_PD-L1_cps) were considered separately.
Time Frame: Baseline biopsy (BX1) before treatment, end of therapy (EOT) surgery 2nd core biopsy (BX2) 3-7 days following last dose of pre-chemotherapy pembrolizumab (i.e after the second dose of pembrolizumab)
Population: Positive RPB indicates a positive relationship between the BFA pCR and continuous factor PDL-1-CPS as values of BFA pCR increase, the value of the continuous factor PDL-1-CPS tends to increase. The positive RPB means that pCR patient group tends to have larger PDL-1-CPS score. The negative RPB indicates an inverse relationship between the binary factor pCR and continuous factor PDL-1-cps. The negative RPB indicates pCR patient group tends to have lower PDL-1-cps score.
Measure: Number (95% Confidence Interval); unit: Corr. Coefficient pCR & PD-L1 CPS
Units Other Than Participants: Tumor Biopsies
Arm/Group | Cohort A: Triple Negative Breast Cancer (TNBC) | Cohort B: HER2-negative Hormone Receptor-positive Tumors | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab
Number analyzed (Participants) | 16 | 13 | 6
Number analyzed (Tumor Biopsies) | 32 | 26 | 12
Corr. Coefficient pCR & PD-L1 CPS
  BX2 (only) CPS After Therapy | 0.1211 [-0.3986 to 0.5818] | 0.0031 [-0.5489 to 0.5531] | -0.0094 [-0.8147 to 0.8084]
  Change CPS of BX2-BX1 | 0.44541 [-0.0645 to 0.7709] | -0.4719 [-0.8118 to 0.1068] | -0.8011 [-0.9773 to 0.0299]

10. Secondary Outcome: Change of Intensity of PD-L1 Expression by Assay as it Relates to Pathologic Complete Response pCR Rates From Chemotherapy Tumor Samples for Proprietary PD-L1 Staining.
Description: A semi-quantitative method used to assess the expression level of proteins or other markers in tissue samples, particularly in immunohistochemistry (IHC) studies. It helps to determine the intensity and proportion of staining, providing a numerical representation of biomarker abundance. The H-score is calculated by multiplying the percentage of positive cells by their staining intensity and summing these values, as described in Dolled-Filhart et al, which calculates a score based on intensity of tumor staining and the percentage of cells implemented. Point Biserial correlation coefficient (RPB) was calculated to quantify the association between the binary factor pCR, and continuous factor PDL-1-Hscore.The PD-L1-Hscore variables (BX2_PD-L1_Hscore, Change_PD-L1_Hscore) were considered separately.
Time Frame: Baseline biopsy (BX1) prior to therapy, EOT surgery 2nd core biopsy (BX2) 3-7 days following last dose of pre-chemotherapy pembrolizumab
Population: Positive RPB indicates a positive relationship between the binary factor pCR and continuous factor PDL-1-Hscore. As the binary factor pCR value increases, the value of the continuous factor PDL-1-Hscore also tends to increase. The positive RPB means that pCR patient group tends to have higher PDL-1-Hscore. A negative RPB indicates an inverse relationship between the binary factor pCR and continuous factor PDL-1-Hscore, a negative RPB indicates pCR patient group tends to have lower PDL-1-Hscore.
Measure: Number (95% Confidence Interval); unit: Corr. Coefficient pCR & PD-L1 H-Score
Units Other Than Participants: Tumor Biopsies
Arm/Group | Cohort A: Triple Negative Breast Cancer (TNBC) | Cohort B: HER2-negative Hormone Receptor-positive Tumors | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab
Number analyzed (Participants) | 17 | 14 | 6
Number analyzed (Tumor Biopsies) | 34 | 28 | 12
Corr. Coefficient pCR & PD-L1 H-Score
  BX2 (only) Hscore (After therapy) | 0.25211 [-0.2601 to 0.6535] | 0.7121 [0.2917 to 0.9019] | -0.3647 [-0.9076 to 0.6348]
  Change_Hscore of Bx-2-Bx-1 | 0.3699 [-0.1347 to 0.7221] | -0.1407 [-0.6246 to 0.4213] | -0.8592 [-0.9844 to -0.15734]

11. Secondary Outcome: Evaluation of Myeloid-derived Suppressor Cells (MDSC) Identified in Blood Samples Post-decitabine Compared to MDSC Found in Blood Samples Collected at Baseline.
Description: Evaluate the level of circulating MDSC per ml of blood at baseline, following treatment with decitabine alone.
Time Frame: Assessed at end of administration of decitabine compared to assessment at baseline prior to protocol treatments.
Measure: Mean (Standard Deviation); unit: absolute cell count per ml of blood
Arm/Group | Cohort A: Triple Negative Breast Cancer (TNBC) | Cohort B: HER2-negative Hormone Receptor-positive Tumors | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab
Number analyzed (Participants) | 20 | 18 | 7
absolute cell count per ml of blood
  Baseline Granulocytic | 13271.20 (24742.36) | 22575.50 (34814.99) | 77038.71 (127561.51)
  Post Decitabine- Granulocytic | 6279.00 (8391.41) | 38759.50 (67973.42) | 43120.00 (60999.23)
  Change- Granulocytic | -6992.20 (27388.05) | 16184.00 (46253.09) | -33918.71 (107087.59)
  Baseline- Monocytic | 59222.05 (85757.80) | 45450.33 (46641.67) | 15843.29 (10160.61)
  Post Decitabine- Monocytic | 20524.50 (16081.57) | 18886.00 (18101.69) | 16081.57 (13631.21)
  Change | -38697.55 (77519.71) | -26564.33 (35958.06) | 238.29 (10580.07)
  Baseline- Total-MDSC | 83927.60 (96291.84) | 213321.11 (579434.80) | 138957.43 (222790.89)
  Post Decitabine- Total MDSC | 35606.00 (26267.93) | 146345.39 (310850.15) | 92662.71 (100386.82)
  Change- Total MDSC | -48321.60 (89365.64) | -66975.72 (283701.53) | -46294.71 (146651.36)

12. Secondary Outcome: Evaluation of Myeloid-derived Suppressor Cells (MDSC) Identified in Blood Samples Post-pembrolizumab Compared to MDSC Found in Blood Samples Collected at Baseline.
Description: Evaluate the level of circulating MDSC per ml of blood at baseline, following treatment with decitabine, and following treatment with decitabine and 2 doses of pembrolizumab.
Time Frame: Assessed at baseline, after administration of decitabine, after decitabine and 2 doses of pembrolizumab.
Measure: Mean (Standard Deviation); unit: Absolute cell count per ml of blood
Arm/Group | Cohort A: Triple Negative Breast Cancer (TNBC) | Cohort B: HER2-negative Hormone Receptor-positive Tumors | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab
Number analyzed (Participants) | 20 | 18 | 7
Absolute cell count per ml of blood
  Baseline- Granulocytic | 13271.20 (24742.36) | 22575.50 (34814.99) | 77038.71 (127561.51)
  Post Pembrolizumab- Granulocytic | 33099.40 (83017.97) | 25780.33 (34038.45) | 63045.29 (87400.02)
  Change(Post Pembro-Baseline) Granulocytic | 19828.20 (81974.04) | 3204.83 (38451.35) | -13993.43 (136887.63)
  Baseline- Monocytic | 59222.05 (85757.80) | 45450.33 (46641.67) | 15843.29 (10160.61)
  Post Pembrolizumab- Monocytic | 22499.95 (23347.79) | 21651.56 (38761.10) | 18028.43 (20787.90)
  Change (Post Pembro- Baseline)- Monocytic | -36722.10 (72130.68) | -23798.78 (53965.00) | 2185.14 (21374.82)
  Baseline- Total MDSC | 83927.60 (96291.84) | 213321.11 (579434.80) | 138957.43 (222790.89)
  Post Pembrolizumab- Total MDSC | 74569.75 (119875.91) | 78836.72 (89861.88) | 133082.00 (91911.07)
  Change (Post Pembro-Baseline)- Total MDSC | -9357.85 (82232.70) | -134484.39 (595746.30) | -5875.43 (203496.45)

13. Secondary Outcome: Event Free Survival (EFS) Rate at 12 Months Following the Last Dose of Pembrolizumab.
Description: Number of patients who are alive and have not had disease relapse at 12 months following last dose of pembrolizumab
Time Frame: 12 Months following surgery
Population: Patients who did not have surgery due to disease progression or experienced disease progression before undergoing surgery were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Triple Negative Breast Cancer (TNBC) | Cohort B: HER2-negative Hormone Receptor-positive Tumors | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab
Number analyzed (Participants) | 18 | 16 | 6
Participants
  Had Progression at 12-month after Surgery | 2 | 0 | 0
  No Progression at 12-month after Surgery | 16 | 16 | 6

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from time of study registration until 30 days following the last dose of decitabine, or until another cancer treatment was initiated, or 30 days following surgery, 12- months.
Arm/Group | Cohort A: Triple Negative Breast Cancer (TNBC) | Cohort B: HER2-negative Hormone Receptor-positive Tumors | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 3/21 | 0/18 | 0/7
Serious Adverse Events (participants affected / at risk) | 7/21 | 6/18 | 4/7
Other Adverse Events (participants affected / at risk) | 21/21 | 18/18 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Triple Negative Breast Cancer (TNBC) (N=21) | Cohort B: HER2-negative Hormone Receptor-positive Tumors (N=18) | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab (N=7)
Adrenal Insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Blood and Lymphatic System Disorders- Other (Blood and lymphatic system disorders) | 0 (0) | 2 (5) | 0 (0)
Catheter Related Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Esophageal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1) | 1 (3)
Gallbladder Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
General Disorders and Administration Site Conditions- Other (General disorders) | 1 (1) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (5)
Infections and Infestations- Other (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Lung Infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Lipase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (4)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic Event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vascular Disorders- Other (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Triple Negative Breast Cancer (TNBC) (N=21) | Cohort B: HER2-negative Hormone Receptor-positive Tumors (N=18) | Cohort A2: Triple Negative Breast Cancer (TNBC) With Extended Pembrolizumab (N=7)
Adrenal Insufficiency (Endocrine disorders) | 2 (2) | 3 (3) | 1 (3)
Alanine Aminotransferase Increased (Investigations) | 2 (2) | 1 (2) | 0 (0)
Alkaline Phosphatase Increased (Investigations) | 2 (2) | 2 (2) | 1 (2)
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 10 (12) | 7 (7) | 4 (7)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Asparate Aminotransferase Increased (Investigations) | 3 (5) | 2 (4) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1)
Cardiac Disorders-Other (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Catheter Related Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholesterol High (Investigations) | 0 (0) | 1 (1) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Creatinine Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dental Carries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 1 (2) | 1 (2)
Disease Progression (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (5)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Edema Face (General disorders) | 2 (2) | 0 (0) | 0 (0)
Edema Limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Esophageal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 8 (10) | 8 (9) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (2)
Fever (General disorders) | 1 (2) | 1 (1) | 1 (3)
Flu Like Symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gait Disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal Disorders- Other (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
General Disorders Administration Site Conditions (General disorders) | 2 (2) | 0 (0) | 0 (0)
Guillain-Barre Syndrome (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 9 (9) | 3 (4) | 3 (3)
Hot Flashes (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (10) | 2 (2) | 1 (1)
Hypoparathyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (6)
Hypothyroidism (Endocrine disorders) | 2 (2) | 1 (2) | 2 (2)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 1 (1)
Investigations- Other (Investigations) | 2 (2) | 1 (1) | 0 (0)
Lipase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (9) | 5 (5) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle Weakness Right-Sided (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail Changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (6) | 6 (8) | 2 (6)
Neck Edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Nervous System Disorders- Other (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutrophil Count Decreased (Investigations) | 15 (17) | 9 (9) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oral Dysesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (2) | 2 (2) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral Motor Neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 1 (1) | 1 (1) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (3) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 5 (9) | 3 (3) | 1 (1)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Thromboembolic Event (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Urine Discoloration (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vaccination Site Lymphadenopathy (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vaccination Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vaginal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular Disorders- Other (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (6)
Weight Loss (Investigations) | 1 (1) | 1 (1) | 0 (0)
White Blood Cell Decreased (Investigations) | 17 (18) | 13 (14) | 2 (2)

LIMITATIONS AND CAVEATS:
Adequate paired biopsy specimens for Tumor and Stroma With Infiltrating Lymphocytes (TIL) and protein Programmed Death-Ligand 1 (PD-L1) analysis were not obtained for all of the enrolled and treated patients due to insufficient tissue amounts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data and results will be owned by the institution. Subject to the terms and conditions of this agreement, institution and principal investigator have the right to publish or publicly present the results of the study. Merck shall have the right to review and comment on any public presentation. No public presentation shall contain any confidential information of Merck.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT02957968/Prot_SAP_002.pdf
  • Informed Consent Form (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT02957968/ICF_000.pdf